CLINICAL TRIAL: NCT06675019
Title: The Effect of Manual Therapy Versus Kinesio Taping on Tension-type Headache in Jouf University Female Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rokaia Ali Zainelabedeen Mohamed Toson, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-92
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Tension Type Headache
Keywords: tension type headache; manual therapy; kinesio taping
MeSH Terms: conditions — Tension-Type Headache | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual therapy (Experimental)
  Interventions: Other: Manual therapy
- Kinesio taping (Experimental)
  Interventions: Other: Kinesio taping
- Control group (Active Comparator)
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Manual therapy — Manual therapy group: will have manual therapy and relaxation training three times per week in addition to their medications as needed. Manual therapy will include stretching exercises, strengthening exercises, soft tissue manipulation in the form of myofascial release and deep friction massage, and postural correction.
  Arms: Manual therapy
Other: Kinesio taping — Kinesio taping group: will have kinesio taping (KT), and relaxation exercises three times per week in addition to their medication as needed, One I-shaped tape was used to apply KT to the upper trapezius muscle that was 50 mm broad and 0.5 mm thick. The tape was measured from the acromion to the hairline in the back, and the upper trapezius fibers were stretched in the extended position, i.e., the cervical vertebrae were flexed to the opposite side and applied to the same side in the flexion and rotation positions. The band was secured to the acromion's insertion site in its first resting position. The muscle was lengthened, and the band was fixed with the initial skin shift, after which the band was fixed to the origin of the hairline from the muscle with a 10% stretch. The tape was massaged with the muscle in the extended position.
  Arms: Kinesio taping
Other: Control (Standard treatment) — The control group will just receive relaxation exercises three times per week, in addition to their medications as needed.
  Arms: Control group

SUMMARY:
Patients suffering from Tension Type Headache (TTH) report emotional and functional deficits (missing work, sleep disorders, emotional stability) and are susceptible to pharmaceutical abuse. Cervical muscle training, posture correction, spinal mobilization, and other physical therapy modalities may help alleviate symptoms.

This study will aim to compare the effect of manual therapy and kinesio taping on tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Students between the ages of 18 and 25 will be enrolled in the study if they have tension type headache based on the IHS headache classification: A headache that occurs at least 15 days per month for more than 3 months (≥ 180 days per year) and lasts for hours or is continuous. The headache exhibits at least one of the following characteristics: 1. bilateral location, 2. pressing/tightening (non-pulsating) character, 3. mild or moderate intensity that is not exacerbated by routine physical activity such as walking or ascending stairs, and both of the following: 1. No more than one of photophobia, phonophobia, or mild nausea, and 2. No moderate to severe nausea or vomiting.

Exclusion Criteria:

* Reumatoid arthritis, suspected malignancy, pregnancy, regular use of triptans, ergotamines, or opioids on ≥ 10 days/month or simple analgesics on ≥ 15 days/month for ≥ 3 months, or physical therapy treatment within 2 months prior to enrollment in the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analouge Scale | 8 weeks
  The Visual Analogue Scale (VAS) will be used to assess the students' headache intensity before the intervention, after one month, and at the end intervention. VAS is used to transform some numerical values, such as pain, to numeric values. The two extremes of a 10 cm line are to be assessed on two extremes, and the patient is requested to indicate where the degree of the pain is appropriate by drawing a line or pointing.

SECONDARY OUTCOMES:
The 6-item headache questionnaire | 8 weeks
  The 6-item headache questionnaire will be examined before the intervention, after one month, and at the end intervention; it comprises six items (pain intensity, social functioning, role functioning, vitality, cognitive functioning, and psychological distress), each with five response alternatives. Never: 6 points, rarely: 8 points, sometimes: 10 points, very frequently: 11 points, and always: 13 points, with a total score ranging from 36 to 78 points.
A headache diary | 8 weeks
  A headache diary will include recording the data at the end of the day to create a record of the clinical history of pain, including frequency, duration (hours per day), headache intensity (Visual Analogue Scale [VAS]: 0-10), and analgesic use.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt